CLINICAL TRIAL: NCT02342327
Title: Smoking Cessation in Menthol Flavored Cigarette Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1406M51364
Record Dates: First submitted 2015-01-14; First posted 2015-01-19 (Estimated); Results first posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continue smoking menthol cigarettes (Other): Menthol cigarette smokers continue to smoke menthol cigarettes for a four week period before attempting to quit smoking
  Interventions: Other: continue smoking menthol cigarettes prior to cessation attempt
- Switch to non-menthol cigarettes (Other): Menthol cigarette smokers switch to non-menthol cigarettes for a four week period before attempting to quit smoking
  Interventions: Other: switch to non-menthol cigarettes prior to cessation attempt

INTERVENTIONS:
Other: switch to non-menthol cigarettes prior to cessation attempt
  Arms: Switch to non-menthol cigarettes
Other: continue smoking menthol cigarettes prior to cessation attempt
  Arms: Continue smoking menthol cigarettes

SUMMARY:
The purpose of this study is to determine if in smokers of menthol cigarettes, switching to non-menthol cigarettes prior to a cessation attempt results in greater cessation success than attempting to quit without first switching

ELIGIBILITY:
Inclusion Criteria:

* Self identify as African American
* smoke primarily menthol cigarettes
* be between the ages of 18 and 64
* smoke a minimum number of cigarettes per day
* express an interest in quitting smoking

Exclusion Criteria:

* current unstable medical / psychiatric condition
* regular use any form of nicotine or tobacco other than cigarettes
* are pregnant or breast feeding

The investigators will evaluate if there are other reasons why someone may not be eligible to participate

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 122 (Actual)
Dates: Start 2014-10-28 (Actual); Primary Completion 2018-07-11 (Actual); Study Completion 2018-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kotlyar, PharmD, Principal Investigator — University of Minnesota
Locations (1):
- Clinical and Translational Sciences Institute, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Kotlyar M, Shanley R, Dufresne SR, Corcoran GA, Okuyemi KS, Mills AM, Hatsukami DK. Effects on Smoking Behavior of Switching Menthol Smokers to Non-menthol Cigarettes. Nicotine Tob Res. 2021 Oct 7;23(11):1921-1927. doi: 10.1093/ntr/ntab090. PMID 33983396
- [Derived] Kotlyar M, Shanley R, Dufresne SR, Corcoran GA, Okuyemi KS, Mills AM, Hatsukami DK. Effects on time to lapse of switching menthol smokers to non-menthol cigarettes prior to a cessation attempt: a pilot study. Tob Control. 2021 Sep;30(5):574-577. doi: 10.1136/tobaccocontrol-2020-055689. Epub 2020 Jul 27. PMID 32719011

RESULTS

PARTICIPANT FLOW:
Groups:
- Continue Smoking Menthol Cigarettes: Menthol cigarette smokers continue to smoke menthol cigarettes for a four week period before attempting to quit smoking
  continue smoking menthol cigarettes prior to cessation attempt
- Switch to Non-menthol Cigarettes: Menthol cigarette smokers switch to non-menthol cigarettes for a four week period before attempting to quit smoking
  switch to non-menthol cigarettes prior to cessation attempt
Period: Overall Study
Arm/Group | Continue Smoking Menthol Cigarettes | Switch to Non-menthol Cigarettes
Started | 60 | 62
Completed Quit Day Visit | 54 | 53
Completed | 39 | 40
Not Completed | 21 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Continue Smoking Menthol Cigarettes | Switch to Non-menthol Cigarettes | Total
Number analyzed (Participants) | 60 | 62 | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (10) | 45 (11) | 46 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 23 | 45
  Male | 38 | 39 | 77
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 60 | 62 | 122
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 60 | 62 | 122

OUTCOME MEASURES:

1. Primary Outcome: Time to Lapse
Description: Time from smoking cessation until first lapse (i.e. a cigarette is smoked)
Time Frame: 6 months
Population: Participants who attended the quit day visit
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Continue Smoking Menthol Cigarettes | Switch to Non-menthol Cigarettes
Number analyzed (Participants) | 54 | 53
days | 1.07 [0.94 to 2.70] | 2.55 [1.65 to 4.46]
Statistical Analysis 1: Comparison: Continue Smoking Menthol Cigarettes; Hazard ratio for time to lapse to smoking in the group switched to non-menthol cigarettes relative to the group continuing to smoke menthol cigarettes; Test type: Other; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.55 to 1.22]

2. Secondary Outcome: Time to Relapse
Description: Days from the quit attempt until the first of seven consecutive smoking days
Time Frame: 6 months
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Continue Smoking Menthol Cigarettes | Switch to Non-menthol Cigarettes
Number analyzed (Participants) | 54 | 53
days | 7 [2 to 32] | 42 [10 to 84]
Statistical Analysis 1: Comparison: Continue Smoking Menthol Cigarettes; Hazard ratio for time to relapse to smoking in the group switched to non-menthol cigarettes relative to the group continuing to smoke menthol cigarettes; Test type: Other; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.42 to 1.06]

ADVERSE EVENTS:
Time Frame: For the duration of each participant's participation (up to 7 months for each participant)
Arm/Group | Continue Smoking Menthol Cigarettes | Switch to Non-menthol Cigarettes
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/62
Other Adverse Events (participants affected / at risk) | 0/60 | 0/62

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-26): https://cdn.clinicaltrials.gov/large-docs/27/NCT02342327/Prot_SAP_000.pdf